CLINICAL TRIAL: NCT06850922
Title: A Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of RO7446603 Administered Alone or in Combination With Aflibercept or Faricimab in Patients With Diabetic Macular Edema
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of RO7446603 Administered Alone or in Combination With Aflibercept or Faricimab in Participants With Diabetic Macular Edema
Acronym: THAMES
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR43828; ISRCTN14152148 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2025-02-26; First posted 2025-02-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept; faricimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Phase 1 segment of this study was open-label and participants were randomized in Part 4. The Phase 2 segment will be a randomized, double-blinded study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Single Ascending Dose (SAD) Stage (Experimental): Participants received a single dose of RO7446603 at five different dose levels as IVT injection on Day 1.
  Interventions: Drug: RO7446603
- Part 2: Multiple Dose (MD) Monotherapy Stage (Experimental): Participants received four different dose levels of RO7446603 (two doses at each planned dose level) as IVT injection, every 8 weeks (Q8W).
  Interventions: Drug: RO7446603
- Part 3: MD Co-administration With Aflibercept Stage (Experimental): Participants received two different dose levels (two doses at each planned dose level) of RO7446603 as IVT injection, Q8W along with four doses of aflibercept IVT injections, every 4 weeks (Q4W).
  Interventions: Drug: RO7446603; Drug: Aflibercept
- Part 4: MD Co-administration With Faricimab Stage (Experimental): Participants received a single dose of faricimab followed by a 4-week enrichment screening period. Eligible participants received two different dose levels (two doses at each planned dose level) of RO7446603 as IVT injection, Q8W, along with three doses of faricimab (co-administered with RO7446603 or alone) as IVT injection, Q4W.
  Interventions: Drug: RO7446603; Drug: Faricimab
- Part 5: MD Co-mixed With Faricimab Stage (Experimental): Participants will receive two different dose levels of RO7446603 (co-mixed with faricimab or faricimab alone) as IVT injection, Q4W for the first six doses followed by Q8W for four doses.
  Interventions: Drug: RO7446603; Drug: Faricimab

INTERVENTIONS:
Drug: RO7446603 — Participants will receive RO7446603 as an IVT injection per the schedule described in the treatment arms.
Drug: Aflibercept — Participants will receive aflibercept as an IVT injection per the schedule described in the treatment arm.
  Arms: Part 3: MD Co-administration With Aflibercept Stage
Drug: Faricimab — Participants will receive faricimab as an IVT injection per the schedule described in the treatment arms.
  Other Names: Vabysmo
  Arms: Part 4: MD Co-administration With Faricimab Stage; Part 5: MD Co-mixed With Faricimab Stage

SUMMARY:
This study aims to evaluate the ocular and systemic safety, tolerability and efficacy of RO7446603 in participants with diabetic macular edema (DME). The study consists of 2 segments: Phase I (Parts 1-4) and Phase II (Part 5). Phase I investigated the safety of RO7446603 following a single and multiple intravitreal (IVT) doses as monotherapy or co-administered with IVT aflibercept or IVT faricimab (in separate injections). Phase II will investigate the safety, tolerability, pharmacokinetics (PK) and efficacy of two dose levels of RO7446603 in combination with faricimab, with the two drugs co-mixed and administered as a single IVT injection, compared to faricimab alone. The first participant was enrolled in the Phase I segment on June 22, 2022. Phase I has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of diabetes mellitus (DM) (Type 1 or Type 2) with glycated hemoglobin (HbA1c) < 12%
* Macular thickening secondary to DME involving the center of the fovea > 325 microns
* Decreased VA attributable primarily to DME between 25 and 73 ETDRS letters

Exclusion Criteria:

* Currently untreated DM or previously untreated participants who initiated oral anti-diabetic medication or insulin within 90 days prior to Day 1
* Uncontrolled blood pressure (BP)
* Pregnancy or breastfeeding, or intention to become pregnant during the study
* For Parts 1-4: IVT anti-VEGF treatment within 90 days prior to Day 1; For Part 5: IVT anti-VEGF treatment within 120 days prior to Day 1 or IVT anti-VEGF treatment prior to Day 1 for treatment naïve participants
* Treatment with SUSVIMOTM (ranibizumab injection) prior to Day 1
* Any IVT or periocular (sub-tenons) corticosteroid treatment within 6 months prior to Day 1
* Any current or history of ocular disease other than DME that may confound assessment of the macula or affect central vision
* Proliferative diabetic retinopathy (PDR) in the study eye
* Active or history of uveitis, vitritis (grade trace or above), and/or scleritis in either eye Other protocol-specified inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Parts 1-5: Percentage of Participants With Adverse Events (AEs) | From study start through end of study (Up to approximately 58 months)
Parts 1-5: Percentage of Participants With Ocular AEs | From study start through end of study (Up to approximately 58 months)
Part 1: Change in Best Corrected Visual Acuity (BCVA) Over Time | From Baseline up to Week 16
  BCVA will be measured via Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters using a set of three precision VisionTM or lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified visual acuity (VA) examiner. The range of EDTRS is 0 to 100 letters. Higher scores indicate improvement in VA.
Parts 2-4: Change in BCVA Over Time | From Baseline up to Week 28
  BCVA will be measured via ETDRS chart at a starting distance of 4 meters using a set of three precision VisionTM or lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified VA examiner. The range of EDTRS is 0 to 100 letters. Higher scores indicate improvement in VA.
Part 5: Change From Baseline in BCVA Averaged Over Weeks 52 and 56 | From Baseline up to Week 56
  BCVA will be measured via ETDRS chart at a starting distance of 4 meters using a set of three precision VisionTM or lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified VA examiner. The range of EDTRS is 0 to 100 letters. Higher scores indicate improvement in VA.

SECONDARY OUTCOMES:
Part 5: Proportion of Participants Gaining ≥ 15 Letters in BCVA From Baseline Averaged Over Weeks 52 and 56 | From Baseline up to Week 56
  BCVA will be measured via ETDRS chart at a starting distance of 4 meters using a set of three precision VisionTM or lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified VA examiner. The range of EDTRS is 0 to 100 letters. Higher scores indicate improvement in VA.
Part 5: Percentage of Participants Gaining ≥ 15, ≥ 10, ≥ 5, or ≥ 0 Letters in BCVA From Baseline Over Time | From Baseline up to Week 56
  BCVA will be measured via ETDRS chart at a starting distance of 4 meters using a set of three precision VisionTM or lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified VA examiner. The range of EDTRS is 0 to 100 letters. Higher scores indicate improvement in VA.
Part 5: Percentage of Participants Avoiding a Loss of ≥ 15, ≥ 10, ≥ 5, or ≥ 0 Letters in BCVA From Baseline Over Time | From Baseline up to Week 56
  BCVA will be measured via ETDRS chart at a starting distance of 4 meters using a set of three precision VisionTM or lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified VA examiner. The range of EDTRS is 0 to 100 letters. Higher scores indicate improvement in VA.
Part 5: Change From Baseline in BCVA Score Over Time | From Baseline up to Week 56
  BCVA will be measured via ETDRS chart at a starting distance of 4 meters using a set of three precision VisionTM or lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R) prior to dilating eyes by a trained and certified VA examiner. The range of EDTRS is 0 to 100 letters. Higher scores indicate improvement in VA.
Parts 1-4: Serum Concentration of RO7446603 Total Fab | Part 1: From Baseline up to Week 16; Parts 2-4: From Baseline up to Week 28
Parts 1-5: Aqueous Humor Concentration of RO7446603 Measured as Total Fab | From study start through end of study (Up to approximately 58 months)
Parts 1-5: Number of Participants With Serum Treatment-emergent Anti-drug Antibody (ADA) Formation to RO7446603 | From study start through end of study (Up to approximately 58 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (77):
- United States (70):
  - Barnet Dulaney Perkins Eye Center, Phoenix, Arizona
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Associated Retinal Consultants PC, Phoenix, Arizona
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retinal Diagnostic Center, Campbell, California
  - The Retina Partners, Encino, California
  - Retina Consultants of Orange County, Fullerton, California
  - Retinal Consultants Medical Group, Modesto, California
  - Northern California Retina-Vitreous Associates, Mountain View, California
  - Retinal Consultants Medical Group, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Macula Retina Vitreous Research Institute, Torrance, California
  - University of Colorado - Eye Center - PPDS, Aurora, Colorado
  - Retina Consultants of Southern Colorado PC, Colorado Springs, Colorado
  - Retina Specialists of Colorado, Denver, Colorado
  - Advanced Vision Research Institute, Longmont, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Blue Ocean Clinical Research, Clearwater, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Retina Institute, Jacksonville, Florida
  - Retina Associates of Florida;Retina Associates of Florida, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - Illinois Eye and Ear Infirmary, Chicago, Illinois
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Raj K. Maturi, MD PC, Indianapolis, Indiana
  - The Retina Care Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Chesapeake Retina Centers - Waldorf, Waldorf, Maryland
  - Associated Retinal Consultants - Royal Oak, Royal Oak, Michigan
  - Retina Consultants Minnesota, Saint Louis Park, Minnesota
  - Long Island Vitreoretinal Consultants;Opthalmology, Hauppauge, New York
  - Retina Vitreous Surgeons of CNY PC, Liverpool, New York
  - Opthalmic Consultants of LI, Lynbrook, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - North Carolina Retina Associates, Cary, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Graystone Eye, Hickory, North Carolina
  - North Carolina (NC) Retina Associates - Wake Forest Office, Wake Forest, North Carolina
  - Piedmont Retina Specialists, Winston-Salem, North Carolina
  - Cincinnati Eye Institute, Blue Ash, Ohio
  - Ohio State Eye and Ear Institute, Columbus, Ohio
  - Tulsa Retina Consultants, Tulsa, Oklahoma
  - Cascade Medical Research Institute LLC, Springfield, Oregon
  - Erie Retina Research, Erie, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Sewickely Eye Group, Sewickley, Pennsylvania
  - Palmetto Retina Center, West Columbia, South Carolina
  - Charles Retina Institute, Germantown, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Retina & Vitreous of Texas, Bellaire, Texas
  - Texas Retina Associates, Dallas, Texas
  - Valley Retina Institute P.A., McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Consultants of Texas - San Antonio, San Antonio, Texas
  - Brown Retina Institute, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Associates of Utah, PLLC;Clinical Research, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Kapoor Institute, Norfolk, Virginia
  - Virginia Eye Institute - Richmond - 7301 Forest Ave, Richmond, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington
- China (6):
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality
  - Eye Hospital,WMU(Zhejiang Eye Hospital), Wenzhou, Zhejiang
  - Beijing Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Shanghai General Hospital - North Campus, Shanghai
- Emanuelli Research and Development Center LLC, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing